CLINICAL TRIAL: NCT00229905
Title: A Case Report of a Child With Anomalous Drainage of the Inferior Vena Cava to the Left Atrium
Brief Title: Child With Anomalous Drainage of IVC to Left Atrium
Status: Terminated | Type: Observational
Why Stopped: sufficient data
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-042
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric health; children; single case study
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to see if any conclusions can be drawn about the uncommon heart defect: anomalous drainage of the inferior vena cava to the left atrium.

DETAILED DESCRIPTION:
Dr. Kogon would like to do a case-report and review of the literature regarding children with the diagnosis of anomalous drainage of the inferior vena cava to the left atrium. At Children's Healthcare of Atlanta, we have seen a single patient with this diagnosis in 2004 and Dr. Kogon would like to discuss this patient in combination with the others already in the literature to see if any conclusions can be drawn about this uncommon heart defect. Currently there are about 20 cases reported in the literature and Dr. Kogon will be reporting on this one case seen in 2004.

The case report of our patient will utilize his medical chart. We hope to provide a brief summary of his clinical presentation, his radiographic evaluation, his operative findings, and his outcome. The only PHI that will be collected will be dates (i.e. date of birth, dates of procedures).

ELIGIBILITY:
Inclusion Criteria:

* single case
* child with anomalous drainage of the inferior vena cava to the left atrium
* at Children's Healthcare of Atlanta

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: child with anomalous drainage of the inferior vena cava to the left atrium
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-03; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States